CLINICAL TRIAL: NCT03527394
Title: The Readiness and Motivation Interview for Families (RMI-Family) Managing Pediatric Obesity
Brief Title: Motivation to Change Lifestyle Habits in Youth With Obesity
Acronym: RMI-Family
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Pro00051447
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Pediatric Obesity; Motivational Interviewing
Keywords: Obesity; Pediatric; Parent; Family; Motivational Interviewing; Lifestyle; Health Behavior
MeSH Terms: conditions — Pediatric Obesity; Obesity; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Families: We plan to recruit a sample of 100 families (dyads) for this study, which will include 100 youth and 100 parents.
  Note: For the sake of transparency, this sample size differs from the original estimate (n=250 families; see Ball et al., BMC Health Serv Res, 2017;17:261). A recent systematic review (Park et al., Int J Nurs Stud, 2018;79:58-69) suggested that sample size estimates for studies that evaluate test-retest reliability (a key psychometric property we will examine) should include ~5 participants for every survey item. Given the design of the interview, and in light of current patient volumes at the clinical recruitment sites, we are confident that a sample of 100 families will be both achievable and satisfactory for psychometric analyses.

SUMMARY:
Approximately one-third of Canadian children have excess weight, putting them at increased risk of type 2 diabetes, cardiovascular disease, bone and joint problems, and some forms of cancer. Because current therapies for managing obesity have modest success, there is a need to develop and test innovative strategies to enhance pediatric weight management. Using a novel interview designed to measure motivation to change lifestyle habits, interviewers will conduct separate and structured 1-on-1 interviews with youth with obesity and parents. By applying principles of motivational interviewing, trained interviewers will ask youth and their parents about their motivation to change lifestyle habits related to diet and physical activity. Subsequently, interview data will be used to examine predictors of clinically-meaningful outcomes over time, including changes in weight status, lifestyle habits, health care utilization, and attrition. The investigators will also measure a number of variables related to weight management, including dietary intake, physical activity, anthropometry, and psychosocial health.

DETAILED DESCRIPTION:
The Readiness and Motivation Interview for Families (RMI-Family) was created as a structured interview for assessing youth and parent motivation (and within family member agreement) regarding lifestyle changes in pediatric weight management.

The RMI-Family was modeled on the Readiness and Motivation Interview (RMI), which was developed originally for use in the management of eating disorders (e.g., anorexia nervosa) and emerged as a 'gold standard' approach to assessing treatment motivation in that population. The RMI-Family was based on the tenets of motivational interviewing (MI), a directive, client-centered, and empirically-supported clinical approach to helping individuals resolve ambivalence about change across a range of lifestyle behaviours, including smoking, substance abuse, as well as diet and physical activity.

Participants will be recruited and enrolled into the study after being referred for pediatric weight management within Alberta Health Services, the governmental authority responsible for providing health care in the province of Alberta, Canada. Interviews will be completed following referral and before youth and parents initiative pediatric weight management. Each youth and parent will complete the RMI-Family (interview duration: 60 - 90 minutes) at baseline, 6-, and 12-months post-baseline. Individual (i.e., youth or parent) and family-level (i.e., across youth and parent) responses to interview questions will be scored, as will aspects of interview administration (e.g., fidelity to motivational interviewing tenets).

Families (youth+parent) will also complete the following questionnaires at baseline, 6- and 12-months follow-up:

1. Behavior Assessment System for Children-Third Edition (BASC-3)
2. Behavior Rating Inventory of Executive Function-Second Edition (BRIEF 2)
3. Emotion Regulation Questionnaire (ERQ)
4. Coping with Children's Negative Response Scale (CCNES)
5. Marlowe-Crowne Social Desirability Scale (MC-SDS)
6. Motivation to Change Rulers (Readiness to change lifestyle habits)
7. Waterloo Eating Behaviour Questionnaire (WEB-Q)
8. Dutch Eating Behaviour Questionnaire (DEBQ)

Physical activity will be measured for youth over a 7-day period using accelerometry, which will provide estimates of total movement time (and movement intensity) and sleep. Data regarding demography (e.g., gender, date of birth), anthropometry (e.g., height, weight), health services utilization (e.g., number of clinic appointments, length of appointments), and program attrition will be retrieved from medical records.

To ensure research team members who administer the RMI-Family interview adhere to principles of motivational interviewing (MI) (e.g., express and show empathy, roll with resistance, support autonomy, take curious and non-judgmental approach), the investigators implemented a number of training procedures before the study launched in fall, 2017. First, as background, all interviewers received and reviewed a package of information and resources (including sample videos) regarding MI, which covered a range of theoretical and practical issues. Second, all interviewers completed practice interviews using the RMI-Family with friends or colleagues that were audio-recorded for their own practice and self-reflection. Third, interviewers completed and audio-recorded 2 - 3 formal interviews (youth and parent versions), which were subsequently reviewed and evaluated by senior research team members with advanced training and expertise in psychology, counseling, and MI. Interviewers received feedback (both positive and constructive) about their interviews; when deemed necessary, interviewers completed additional interviews to build competence and skill, which were also reviewed by senior team members until they were confident that a similar and high level of proficiency was achieved by all interviewers.

To ensure interviewers maintain a high level of competence in administering the RMI-Family interview, all youth and parent interviews will be recorded (audio only) over the course of this study. After each interviewer completes 5 interviews, he/she will submit a randomly-selected interview for review by research team members to ensure implementation fidelity. To assess fidelity, the investigators will use the Motivational Interviewing Supervision and Training Scale (MISTS), which provides a behavioural count of interviewers' skills consistent with the principles of MI and assess the quality and fidelity with which the interview is administered. Subsequently, interviewers and reviewers will discuss issues related to clinical interactions and conversations; this formative approach is designed to optimize adherence to the MI interviewing practices over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years old
* Youth with an age- and sex-specific BMI ≥97th percentile.
* Parents or guardians who self-identify as the primary caregiver of the youth and are able to provide in-depth perspective on youth lifestyle habits.
* Youth and parents who are proficient in English (reading and communicating).

Exclusion Criteria:

* <13 or >18 years old
* Youth with an age- and sex-specific BMI <97th percentile.
* Parents or guardians who do not self-identify as the youth primary caregiver or are not able to provide in-depth perspective on youth lifestyle habits.
* Families who are not proficient in English (reading and communicating).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Youth with obesity (BMI ≥97th percentile) and their parents. The study will be conducted at multiple sites within Alberta Health Services, including those families referred to and enrolled in multidisciplinary weight management clinics (Pediatric Centre for Weight and Health [PCWH]) at the Stollery Children's Hospital (Edmonton, AB) and Alberta Children's Hospital (Calgary, AB) and outpatient nutrition counseling for pediatric weight management (Edmonton, AB). The outpatient nutrition counseling occurs within clinic space at the PCWH in Edmonton, AB.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline psychometric properties at 6- and 12-months | Baseline, 6- and 12-months post-baseline
  A number of psychometric properties of the Readiness and Motivation Interview for Families (RMI-Family) will be examined, including internal consistency, test-retest reliability, convergent validity, and concurrent validity. Based on data derived from the RMI-Family, we will generate youth, parent, and family (youth-parent) total motivation and motivation sub-scores (5-point Likert scale).

SECONDARY OUTCOMES:
Predictive value of the Readiness and Motivation Interview (RMI-Family) | Baseline, 6- and 12-months post-baseline
  Predictive validity of the RMI-Family will be examined by relating youth, parent, and family (youth-parent) scores (5-point Likert scale) from the interview to clinically-meaningful outcomes at baseline, 6- and 12-month follow-up, including anthropometry, lifestyle habits, psychosocial health, health care use, and program attrition.

CONTACTS AND LOCATIONS:
Overall Officials: Geoff DC Ball, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Alberta Children's Hospital (Pediatric Centre for Weight and Health), Calgary, Alberta
  - Stollery Children's Hospital (Pediatric Centre for Weight and Health), Edmonton, Alberta

REFERENCES:
- [Background] Geller J, Avis J, Srikameswaran S, Zelichowska J, Dartnell K, Scheuerman B, Perez A, Rasquinha A, Brown KE, Chanoine JP, Ball G. Developing and Pilot Testing the Readiness and Motivation Interview for Families in Pediatric Weight Management. Can J Diet Pract Res. 2015 Dec;76(4):190-3. doi: 10.3148/cjdpr-2015-024. Epub 2015 Aug 17. PMID 26280565
- [Background] Ball GD, Spence ND, Browne NE, O'Connor K, Srikameswaran S, Zelichowska J, Ho J, Gokiert R, Masse LC, Carson V, Morrison KM, Kuk JL, Holt NL, Kebbe M, Gehring ND, Cesar M, Virtanen H, Geller J. The readiness and motivation interview for families (RMI-Family) managing pediatric obesity: study protocol. BMC Health Serv Res. 2017 Apr 11;17(1):261. doi: 10.1186/s12913-017-2201-8. PMID 28399913
- See also: The Readiness and Motivation Interview for Families (RMI-Family) Managing Pediatric Obesity: study protocol — https://bmchealthservres.biomedcentral.com/track/pdf/10.1186/s12913-017-2201-8?site=bmchealthservres.biomedcentral.com